CLINICAL TRIAL: NCT07102056
Title: Prospective Study of 18F-AlF-NOTA-Octreotide PET-CT or PET-MR in Diagnosis, Treatment and Prognosis for Neuroendocrine Neoplasms
Brief Title: 18F-AlF-NOTA-Octreotide PET in Neuroendocrine Neoplasms
Status: Not yet recruiting | Type: Observational
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: FirstZhejiangU-18OC-NENs
Record Dates: First submitted 2025-07-08; First posted 2025-08-03 (Actual); Last update posted 2025-12-29 (Actual); Status verified 2024-12

CONDITIONS: Neuroendocrine Tumors
MeSH Terms: conditions — Neuroendocrine Tumors

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

INTERVENTIONS:
Diagnostic Test: 18F-AlF-NOTA-Octreotide PET-CT or PET-MR — 18F-Octreotide PET/CT or PET/MR And enhanced CT or MR Imaging

SUMMARY:
The study aims to elucidate how 18F-Octreotide PET/CT or PET-MR can assist in accurate localization, treatment planning, prognostic predictions, and the selection of PRRT efficacy in neuroendocrine tumors. It also highlights important applications in lesion segmentation measurement, tumor grading, prognostic survival prediction, and genotype identification.

ELIGIBILITY:
Inclusion Criteria:

1. Clinical diagnosed of neuroendocrine neoplasms.
2. Suspected of neuroendocrine neoplasms.

Exclusion Criteria:

1. Inability to undergo biopsy/surgical treatment.
2. Concurrent active malignancy.
3. Severe uncontrolled comorbidities/active infections.
4. Inability to provide informed consent.

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a previous diagnosis of neuroendocrine tumors who are suspected of recurrence or metastasis.
Sampling Method: Probability Sample
Enrollment: 152 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-06-03 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic efficacy | through study completion, an average of 1.5 year
  Sensitivity, specificity, positive and negative predictive value of 18F-OC PET/CT and PET/MR Imaging in neuroendocrine neoplasms

OTHER OUTCOMES:
Prognostic Value of Baseline 18F-OC PET for Progression-Free Survival (PFS) in High-Risk Patients | through study completion, 3-4 years
  This measure evaluates the association between baseline 18F-OC PET parameters (e.g., SUVmax, SUVmean, metabolic tumor volume [MTV], total lesion glycolysis [TLG]) and progression-free survival (PFS) in high-risk neuroendocrine neoplasms patients. PFS will be defined as the time from diagnosis to disease progression or relapse, assessed using the Kaplan-Meier method and Cox proportional hazards model.

DOCUMENTS (1):
  • Study Protocol and Informed Consent Form (2024-11-16): https://cdn.clinicaltrials.gov/large-docs/56/NCT07102056/Prot_ICF_000.pdf